CLINICAL TRIAL: NCT02834572
Title: Using Technology to Match Young Black Men and Transwomen Who Have Sex With Men or Transwomen to HIV Testing Options
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: New York Blood Center (Other)
Responsible Party: Principal Investigator, Beryl Koblin, Ph, D., Principal Investigator, New York Blood Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 473699-41
Record Dates: First submitted 2016-05-23; First posted 2016-07-15 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: HIV Testing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- All About Me (Experimental): assessment and algorithm to provide participants with a tailored recommendation of their optimal HIV testing approach
  Interventions: Behavioral: All About Me
- Control (Active Comparator): HIV testing information
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: All About Me — Assessment and algorithm to determine recommended HIV testing approach
  Arms: All About Me
Behavioral: Control — HIV testing information
  Arms: Control

SUMMARY:
Young Black men who have sex with men (MSM) and transwomen in the US are affected by HIV at severely disproportionate rates. A key component of HIV prevention for communities at risk is diagnosing HIV infections through regular HIV testing. A significant proportion of young Black MSM and transwomen have not tested in the prior year. This research study seeks to address low HIV testing rates among young Black MSM and transwomen by testing a brief Internet-based HIV testing intervention optimized for mobile devices. The intervention takes advantage of the variety of HIV testing options now available, including the HIV self testing, couples-based HIV counseling and testing and traditional clinic-based testing and will provide men and transwomen with a tailored recommendation of their optimal HIV testing approach. The investigators are conducting a pilot randomized study among young Black MSM and transwomen followed for 6 months to estimate the intervention's potential efficacy in increasing HIV testing.

DETAILED DESCRIPTION:
We are conducting a pilot study among 240 young Black MSM and transgender women randomized to the Intervention Arm (assessment and algorithm to deliver a tailored recommendation) or Control (assessment and standard HIV testing information) and followed for 6 months to estimate the intervention's potential efficacy in increasing HIV testing. After informed consent, participants are asked to provide contact information on the locator form. Then, participants complete a brief quantitative assessment including basic demographics, HIV testing history and other factors related to HIV testing. All participants, regardless of study arm, then receive information about each HIV testing method including how the tests are conducted (blood, oral sample), and availability of counseling and support. Participants then are randomized into 1 of the 2 study arms. A computer program will randomly assign each participant using randomly ordered block sizes of 4 and 6 and stratified by age (16-23, 24-29 years) to balance groups.

Participants assigned to the Intervention Arm will complete a brief quantitative assessment lasting approximately 2-3 minutes to assess those factors associated with HIV testing and thus are needed to complete the algorithm. They then receive the results of the HIV testing algorithm, presented as their personalized HIV testing approach. All participants will receive information on resources in New York City to test by all of these methods. The control participants are provided with the above information about each testing approach but without a recommended approach.

ELIGIBILITY:
Inclusion Criteria:

* male at birth;
* self-identify as Black, African American, Caribbean Black, African Black or multiethnic Black;
* able to read and respond in English;
* between 16-29 years of age;
* known to be HIV-infected;
* insertive or receptive anal intercourse with a man or transwoman in the last 12 months;
* reside in the New York City metropolitan area

Exclusion Criteria:

* enrolled in any other HIV research study involving HIV testing
* participant in an HIV vaccine trial
* currently taking pre-exposure prophylaxis

Ages: 16 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 236 (Actual)
Dates: Start 2016-06; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants reporting having an HIV test as assessed by questionnaire | 3 months
  Self-reported HIV test in the prior 3 months assessed by questionnaire

SECONDARY OUTCOMES:
Number of participants who are aware of HIV self-testing and couples based voluntary counseling and testing as assessed by questionnaire | 3 months
  Self-reported awareness of HIV self-testing and couples based voluntary counseling and testing assessed by questionnaire
Number of intervention participants recommended a self-test who use a self-test as assessed by questionnaire | 3 months
  Self-reported use of self test among those recommended a self test - Intervention participants only
Number of intervention participants recommended testing at a clinic who test at a clinic as assessed by questionnaire | 3 months
  Self-reported use of testing at a clinic among those recommended to test at a clinic - Intervention participants
Number of intervention participants recommended couples testing who test using couples testing as assessed by questionnaire | 3 months
  Self-reported use of couples testing among those recommended to test using couples testing - Intervention only

CONTACTS AND LOCATIONS:
Overall Officials: Beryl Koblin, PhD, Principal Investigator — NY Blood Center
Locations (1):
- New York Blood Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Frye V, Nandi V, Hirshfield S, Chiasson MA, Wilton L, Usher D, Hoover DR, Koblin BA. Brief Report: Randomized Controlled Trial of an Intervention to Match Young Black Men and Transwomen Who Have Sex With Men or Transwomen to HIV Testing Options in New York City (All About Me). J Acquir Immune Defic Syndr. 2020 Jan 1;83(1):31-36. doi: 10.1097/QAI.0000000000002223. PMID 31809359
- [Derived] Koblin B, Hirshfield S, Chiasson MA, Wilton L, Usher D, Nandi V, Hoover DR, Frye V. Intervention to Match Young Black Men and Transwomen Who Have Sex With Men or Transwomen to HIV Testing Options (All About Me): Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2017 Dec 19;6(12):e254. doi: 10.2196/resprot.8856. PMID 29258976